CLINICAL TRIAL: NCT00671879
Title: Randomized, Double-Blind, Double-Dummy Trial of Two Sustained Release Formulations of Carisoprodol Compared to Placebo in Subjects With Acute, Painful, Musculoskeletal Spasm of the Lower Back
Brief Title: Study to Evaluate Two Formulations of Carisoprodol in Subjects With Musculoskeletal Spasm of the Lower Back
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP511
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Carisoprodol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carisprodol SR 700 mg (Experimental): Carisoprodol 700 mg twice daily
  Interventions: Drug: Carisoprodol SR 700 mg
- Carisoprodol SR 500mg (Experimental): Carisoprodol SR 500 mg twice daily
  Interventions: Drug: Carisoprodol SR 500 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carisoprodol SR 700 mg — 700 mg twice daily tablet
  Other Names: no other name
  Arms: Carisprodol SR 700 mg
Drug: Carisoprodol SR 500 mg — carisoprodol SR 500 mg tablet
  Other Names: no other name
  Arms: Carisoprodol SR 500mg
Drug: Placebo — placebo tablet
  Other Names: no other name
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if two sustained released formulations of carisoprodol are more effective than placebo.

DETAILED DESCRIPTION:
Methodology:

This will be a randomized, double-blind, double-dummy, placebo-controlled, parallel-group study in subjects 18-70 years of age with acute, painful, muscle spasm of the lower back. The study consists of a baseline screening (Study Day 1), during which subjects will be evaluated for inclusion/exclusion criteria, and a 7-day double-blind treatment period (Study Day 1 through Study Day 7). Subjects will be randomly assigned to be dosed twice daily with one of the following double-blind treatments: SR carisoprodol 500-mg tablets, SR carisoprodol 700-mg tablets, or placebo.

Subjects will be evaluated in the clinic on Study Days 1, 3 and 7. Subjects who remain symptomatic on Study Day 7 will be allowed to continue in the study for a 7-day, double-blind extension period at the discretion of the Investigator. Subjects will be contacted by telephone for a safety follow-up 7 days after the last dose of study medication.

A pharmacokinetic (PK) substudy will be conducted at selected sites. These sites will obtain blood samples for PK analysis at the end of the 7-day treatment period and the 14-day treatment period, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Onset of pain is within 3 days of first visit
* Subject rating of pain must be 40 mm or greater on VAS
* Ability to discontinue all analgesics, NSAIDs, and other muscle relaxants
* Willingness to provide written informed consent
* Must be in generally good health

Exclusion Criteria:

* Presence of sciatic pain
* History of clinically significant spine pathology such as herniated nucleus pulpous, spondylolisthesis, spinal stenosis
* Presence of underlying chronic back pain
* Neurological signs and symptoms such as numbness, tingling, foot drop, paresthesia, unexplained constipation, urinary retention or urinary incontinence
* Myocardial infarction within one year of study
* Cancer not in remission or in remission less than one year
* HIV or other immunodeficiency syndromes
* History of osteoporosis or at high risk for vertebral fracture
* Underlying rheumatologic disease such as rheumatoid arthritis, ankylosing spondylitis, etc.
* Presence of active influenza or other viral syndromes
* Morbid obesity (BMI >39)
* Evidence of infection, such as low grade fever or neutrophilia
* Existence of any medical/surgical condition that could interfere with the evaluation of the study medication
* Known history of alcohol or drug abuse
* Injury involving high potential for litigation, including worker's compensation or automobile accidents
* Pregnancy or breast feeding
* Women of child-bearing potential not abstinent or not practicing a medically acceptable method of contraception
* Vertebral body or spinous process, percussive tenderness on physical exam
* Any abnormalities in the following tests of both lower extremities: ankle dorsiflexion strength, great toe dorsiflexion strength, absent or hyperreflexic Achilles or patellar tendor reflexes, abnormal sensory exam in the medial, dorsal or lateral aspect of the foot and positive straight leg raise test
* Urgent medical conditions on comprehensive exam that might indicate a more serious condition should be treated urgently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M. Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (73):
- United States (73):
  - Brookwood Internists, P.C., Birmingham, Alabama
  - Gulf Shores General Practice Center, Gulf Shores, Alabama
  - Simon Williamson Clinic, PC, Hueytown, Alabama
  - Vaugh H Mancha Jr., PC Family Practice, Montgomery, Alabama
  - NextCare Institute for Clinical Research, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Quality of life Medical, LLC, Anaheim, California
  - ICT - Beverly Hills, Beverly Hills, California
  - Lovelace Scientific Resources, Inc., Burbank, California
  - Chrishard Medical Group, Inglewood, California
  - Impact Clinical Trials and Powerplay, Los Angeles, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - San Diego Managed Care Group, San Diego, California
  - Crest Clinical Trials, Inc., Santa Ana, California
  - Santa Barbara Clinical Research Inc., Santa Barbara, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Tampa Bay Medical Research, Clearwater, Florida
  - Atlantic Institute of Clinical Research, Daytona Beach, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Orthopaedic Assoc. of S. Broward, P.A., Hollywood, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Jay Care Medical Center, Lakeland, Florida
  - Innovative Research of West FL, Inc., Largo, Florida
  - Oslar Medical, Inc./ Osler Clinical Research, Melbourne, Florida
  - Homestead Clinical Research, Naranja, Florida
  - Andres Patron, DO, PA, Pembroke Pines, Florida
  - Wilker/Powers Center for Clinical Studies, Saint Cloud, Florida
  - Orlando Rangel, M.D., P.A., Tampa, Florida
  - West Wind'r Research & Development, LLC, Tampa, Florida
  - Palm Beach Research center, West Palm Beach, Florida
  - PMI Health Research Group, Atlanta, Georgia
  - Perimeter Institute for Clinical Research, Inc., Atlanta, Georgia
  - Best Clinical Research, Decatur, Georgia
  - Dupage Family Medicine, Naperville, Illinois
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Bluegrass Orthopaedics & Hand Care Research, Lexington, Kentucky
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Clinical Research Institute, New Orleans, Louisiana
  - Highland Clinic, APMC, Shreveport, Louisiana
  - Waterford Medical Associates, Waterford, Michigan
  - CRC of Jackson, Jackson, Mississippi
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Dr. Meera Dewan PC, Omaha, Nebraska
  - Association of International Professionals, Las Vegas, Nevada
  - ICT - Las Vegas, Las Vegas, Nevada
  - Immedicenter, Bloomfield, New Jersey
  - Land Clinical Studies, West Caldwell, New Jersey
  - Research Across America, New York, New York
  - Odyssey Research, Fargo, North Dakota
  - Parsons Avenue Medical Clinic, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Hillcrest Clinical Research, Oklahoma City, Oklahoma
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Warminster Medical Association, Warminster, Pennsylvania
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Palmetto Family Medicine Center, Pelzer, South Carolina
  - Holston Medical Group, P.C., Kingsport, Tennessee
  - Medical Clinic of North Texas, Arlington, Texas
  - Central Texas Clinical Research, Austin, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - Texas Family Care Clinical Research, Colleyville, Texas
  - Research Across America, Dallas, Texas
  - Georgetown Medical Clinic, Georgetown, Texas
  - F. Adam Kawley, MD PA, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - GSA Research, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Clinical Health Research, LLC, Sugar Land, Texas
  - Holston Medical Group, P.C., Weber City, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo treatment arm
Period: Overall Study
Arm/Group | Carisprodol SR 700 mg | Carisoprodol SR 500mg | Placebo
Started | 281 | 279 | 280
Completed | 281 | 275 | 274
Not Completed | 0 | 4 | 6
Not completed — Withdrawal by Subject | 0 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carisprodol SR 700 mg | Carisoprodol SR 500mg | Placebo | Total
Number analyzed (Participants) | 281 | 279 | 280 | 840
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 279 | 279 | 280 | 838
  >=65 years | 2 | 0 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.35) | 41.6 (11.79) | 41.4 (11.86) | 41.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 145 | 144 | 438
  Male | 132 | 134 | 136 | 402
Region of Enrollment [Number; unit: participants]
  United States | 281 | 279 | 280 | 840

OUTCOME MEASURES:

1. Primary Outcome: Subject Rated Change Relief From Starting Backache of Pain on a 100-point Visual Analog Scale
Description: on a visual analog scale of 0 to 100 millimeters(mm) with 0 being no pain and 100 being maximum pain By measuring the amount of pain before and during treatment done at each visit and recording the difference in mm.During treatment scores were averaged and this average was compared to the baseline value.
Time Frame: baseline to 14 days
Population: intent to treat(ITT) population least square mean(LSMEAN, LSMEAN) diff vs Placebo
Measure: Least Squares Mean (Standard Deviation); unit: mm
Groups:
- Carisprodol SR 700 mg: Carisoprodol SR 700 mg twice daily
Arm/Group | Carisprodol SR 700 mg | Carisoprodol SR 500mg | Placebo
Number analyzed (Participants) | 270 | 271 | 264
mm | 16.4 (1.30) | 15.5 (1.34) | 15.2 (1.32)

2. Secondary Outcome: Subject Functional Assessment Based on the Roland-Morris Disability Questionnaire (RMDQ)
Description: Subject functional assessment based on the Roland-Morris Disability Questionnaire (RMDQ)at day 14.Subjects were asked to read a list of 24 sentences that people have used to describe themselves when they had back pain, and were asked to mark those statements that described their condition that day. The number of marked statements was added. A decrease in the number of marked statements from baseline represented improvement on the RMDQ.
Time Frame: baseline and day +14
Population: Intent to Treat(ITT) population
Measure: Least Squares Mean (Standard Error); unit: marked statements
Arm/Group | Carisprodol SR 700 mg | Carisoprodol SR 500mg | Placebo
Number analyzed (Participants) | 135 | 141 | 142
marked statements | 4.2 (0.64) | 5.0 (0.64) | 4.3 (0.65)

ADVERSE EVENTS:
Arm/Group | Carisprodol SR 700 mg | Carisoprodol SR 500mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/281 | 3/275 | 0/274
Other Adverse Events (participants affected / at risk) | 98/281 | 94/275 | 49/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carisprodol SR 700 mg (N=281) | Carisoprodol SR 500mg (N=275) | Placebo (N=274)
atypical pneumonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
severe influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carisprodol SR 700 mg (N=281) | Carisoprodol SR 500mg (N=275) | Placebo (N=274)
somnolence (Nervous system disorders) | 27 (27) | 38 (38) | 20 (20)
headache (Nervous system disorders) | 12 (12) | 13 (13) | 10 (10)
dizziness (Nervous system disorders) | 11 (11) | 11 (11) | 4 (4)
nausea (Gastrointestinal disorders) | 14 (14) | 7 (7) | 1 (1)
fatigue (General disorders) | 4 (4) | 6 (6) | 2 (2)
increased blood CPK (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 4 (4)
insomnia (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3)
constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
dry mouth (General disorders) | 1 (1) | 4 (4) | 0 (0)
vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Lasegues Test Positive (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
clumsiness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
pain in extremity (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No